CLINICAL TRIAL: NCT02930057
Title: Transforaminal Epidural Steroid Injection in Conjunction With Pulsed Radiofrequency Treatment of the Lumbar Dorsal Root Ganglion for the Management of Chronic Lumbosacral Radicular Pain: a Randomized, Double-blind Trial
Brief Title: Transforaminal Epidural Steroid Injection With Pulsed Radiofrequency for Chronic Lumbosacral Radicular Pain Management
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Vadim Tashlikov, Senior Doctor, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3301-16-SMC
Record Dates: First submitted 2016-10-06; First posted 2016-10-11 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Radicular; Neuropathic, Lumbar, Lumbosacral; Low Back Pain; Back Pain With Radiation
Keywords: lumbar dorsal root ganglion; transforaminal epidural steroid injection; chronic lumbosacral radicular pain; pulsed radiofrequency treatment; betamethasone; dorsal root ganglion
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Betamethasone; Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celestone (Experimental): all patients of the experimental Celestone group will receive transforaminal epidural injection of the solution of 1 cc of Lidocaine 1% with 1 cc of Celestone® Chronodose® around each dorsal root ganglion immediately after the radiofrequency treatment has been performed.
  Interventions: Drug: Celestone; Procedure: pulsed radiofrequency treatment
- Control (Other): all patients of the control group will receive transforaminal epidural injection of the solution of 1 cc of Lidocaine 1% with 1 cc of normal saline around each dorsal root ganglion immediately after the radiofrequency treatment will be performed.
  Interventions: Procedure: pulsed radiofrequency treatment; Drug: Control

INTERVENTIONS:
Drug: Celestone — all of the patients of the experimental Celestone group will receive transforaminal epidural injection of the solution of 1 cc of Lidocaine 1% with 1 cc of Celestone® Chronodose® around each dorsal root ganglion immediately after the radiofrequency treatment has been performed
  Arms: Celestone
Procedure: pulsed radiofrequency treatment — all of the patients who will participate in the study will receive pulsed radiofrequency treatment adjacent to lumbosacral dorsal root ganglion(s).
Drug: Control — all of the patients of the control group will receive transforaminal epidural injection of the solution of 1 cc of Lidocaine 1% with 1 cc of normal saline around each dorsal root ganglion immediately after the radiofrequency treatment will be performed.
  Arms: Control

SUMMARY:
The purpose of this study is to examine the potential changes in levels of pain, quality of life (QoL) and activities of daily living (ADL) observed when transforaminal epidural steroid injection is administered in conjunction with pulsed radiofrequency treatment of the lumbar dorsal root ganglion during the initial 3 months follow-up period. Safety (monitoring side effects) of the treatment is determined.

The study hypothesis is that the application of transforaminal epidural steroid injection (TFESI) in conjunction with pulsed radiofrequency treatment (PRF) treatment of the lumbar dorsal root ganglion would increase the treatment response of PRF and thereby provide a measurable difference in the pain scores, quality of life and activities of daily living for the patients suffering from chronic lumbosacral radicular pain.

DETAILED DESCRIPTION:
The study sample:

120 (one hundred and twenty) patients diagnosed with chronic lumbosacral radicular pain were elected by their pain specialists to undergo pulsed radiofrequency treatment adjacent to lumbosacral dorsal root ganglion(s). A patient with radicular pain affecting more than one segment on one side will be treated for all the involved segments with the same technique and this will be considered a single intervention for the study.

60 (sixty) patients (the experimental Celestone group) undergoing pulsed radiofrequency treatment will receive transforaminal epidural injection of the solution of 1 cc of Lidocaine 1% with 1 cc of Celestone Chronodose around each dorsal root ganglion immediately after the radiofrequency treatment has been performed. 60 (sixty) patients (the control group) undergoing pulsed radiofrequency treatment will receive transforaminal epidural injection of the solution of 1 cc of Lidocaine 1% with 1 cc of normal saline around each dorsal root ganglion immediately after the radiofrequency treatment will be performed.

Randomization and blinding:

Patients will be randomly assigned to the Celestone group (N = 60) or the control group (N = 60). The allocation of patients into either group will be performed using a computer-generated randomization program. Each patient's randomization number will be concealed until the end of the study from both the patients and the outcome assessor, who will be an independent research coordinator at the investigators pain clinic. The patients will be explained that they will not know which medicine they will receive until the study completion.

Procedure:

The study will take place in the Chaim Sheba TelHashomer Medical Center, Ramat Gan, Israel. Participants will be recruited from the hospital's Pain Management outpatient clinic from the patients eligible for the procedure involving pulsed radiofrequency of the lumbosacral dorsal root ganglion. After receiving the hospital's Helsinki approval, the P.I. and/or other designated staff in the department will approach relevant patients (in line with the mentioned inclusion and exclusion criteria), describe the procedure, inform of the possible adverse events and collect informed consent if the patients are interested in participating. Consent will be obtained from the patient during the patient's visit when the option of RF is agreed upon and scheduled for the future.

Eligible patients will not receive any financial reimbursement. It will be stressed to prospective subjects that participation in the research will have no implications on their treatment in the hospital, or the relationship with their current healthcare providers. The patients will be advised that they may unconditionally revoke their consent at any given time during participation without repercussion on future care. For the first month after the procedure, patients will be instructed not to change their previously prescribed analgesic medications. All patients will be made aware of this guideline prior to study participation. After the first month follow-up visit, the prescribed doses of any analgesics will be increased or decreased in regard to the pain intensity of the patient. Patients who will have increments in analgesic medication or who will be elected for alternative treatments will be considered treatment failure. Data collected during the experiment will be kept in a secure location and will be shredded after the project's completion. All information regarding patients treatment both inside and outside of the project will be kept in the utmost of confidentiality, respecting both legal and ethical constraints.

Patients agreeing to participate in the study will come to the pre-operative room of the Pain Department at the designated time. There they will be monitored, initial intensity of the pain (0 to 10) on the numerical rating scale (NRS) will be recorded and pre-operative vital signs assessed (e.g.- blood pressure, heart rate, oxygen saturation). Each patient will complete the Roland Disability Questionnaire and the Oswestry Disability Index score. All syringes with the solutions to be injected by the transforaminal approach will be prepared prior to entering the operating room. After that the patient will enter the operating room to undergo pulsed radiofrequency treatment. The patient will sign consent for the procedure. The patient will be placed in the prone position with a pillow under the lower abdomen to provide an easy transforaminal approach. It will be forbidden to call name or the dose of any medication which will be injected during the procedure except the 1.5cc of Midazolam IV that will be given for light sedation. Fluoroscopy will be used to identify the specific site of the injections and radiofrequency in all cases. After sterile preparation of the needle insertion area, the skin will be infiltrated with 1% Lidocaine, and a 22-gauge, 4-in radiofrequency needle with a 10 mm curved active tip will be advanced under fluoroscopic guidance. Anatomic landmarks will be identified, and the needle will be positioned closely to the dorsal root ganglion under fluoroscopy guidance. The tip of the needle will be placed in the dorsal-cranial quadrant of the intervertebral foramen on the oblique image, and the tip will be positioned between one-third and halfway to the pedicle column on the antero-posterior image. If intravenous uptake will be occurred, the needle will be repositioned until intravenous uptake was absent and an epidural flow pattern was achieved. If intra-arterial, intrathecal, or intradiscal flow will be identified, the procedure was aborted. After confirmation of epidural spread (using a contrast dye) and the radiofrequency needle positioning adjacent to the appropriate dorsal root ganglion, 1 cc of normal saline will be injected to decrease electrical impedance around the radiofrequency needle. Then the stylet will be replaced by the radiofrequency probe and the probe will be connected to the radiofrequency generator. Defining the final position of the radiofrequency probe will require a sensory stimulation (50 Hz) threshold ≤0.5 V, which will create paresthesia corresponding to the existing distribution of the patient's radicular pain. Then in the two groups of patients two cycles of pulsed radiofrequency will be performed at 42°C for 120 seconds. Immediately after the radiofrequency treatment in the Celestone group the solution of 1 cc of Lidocaine 1% with 1 cc of Celestone Chronodose will be injected around each dorsal root ganglion through the radiofrequency needle. In the control group the solution of 1 cc of Lidocaine 1% with 1 cc of normal saline will be injected.

All patients will be treated according to the protocol. If an emergency situation occurs or in case of unblinding, the treatment will be altered and the patients will be considered withdrawn. Such patients will proceed with conservative or interventional management without unblinding. They will also continue their structured exercise program, as other patients do.

After the procedure the patient will be taken to the recovery room in the pain clinic and will be monitored for at least for 30 minutes. Vital signs will be assessed immediately post-op in the recovery room and again after 30 minutes, just prior to discharge.

Requests for additional analgesia (Optalgin, etc) will be assessed. During the 30 minutes following the entry to recovery room the patients will be asked if they are experiencing any of a number of the symptoms used by the list of adverse events and their responses will noted in their records. All the patients will be warned of potentially serious complications requiring immediate evaluation (e.g. progressive weakness). To examine delayed adverse events the patients will be asked to select any of a number of the symptoms used by the list of adverse events for up to 72 hours after the procedure (the patients will be asked to bring the completed lists of the symptoms to their follow up visit in 1 month after a procedure). All patients will be seen at a follow-up appointment with their pain treating physician in the Pain Department of Tel HaShomer in 1, 2 and 3 months following the procedure.

Results:

The baseline characteristics of all participating patients will be collected. Numerical data will include age, height, weight, body mass index, total duration of pain. Categorical data will include sex, diagnosis, coexisting medical conditions such as diabetes and hypertension, target location, and level of the compromised nerve root(s).

A comprehensive review and statistical analysis of data will be conducted at the completion of the study. Changes in pain scores, as reported by the patients via the NRS scores, will be analyzed before the procedure and at 1, 2 and 3 months postprocedure. Changes in ADL and QoL will be measured using the Roland Disability Questionnaire and the Oswestry low back pain disability scales. Both the Roland Disability Questionnaire and the Oswestry scores will be completed by the patients both before the procedure and at 1, 2 and 3 months postprocedure.

Successful pain relief (responders) will be defined as either ≥50% or ≥4-point pain reduction in the NRS; functional success will be defined as either ≥40% reduction in Roland Disability Questionnaire or Oswestry Disability Index scores.

Data analyses will be carried out with the help of a package of statistical programs Win Pepi (the fourth version). Categorical and continuous data comparison, Chi-squared test (Fisher's exact test where necessary) and t test will be performed.

The outcome data of the patients will be measured at 4 periods of time therefore a repeated measures analysis of variance will be performed. A P value of less than 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* age ≥18 years old,
* pain intensity≥4 out of 10 on the numerical rating scale (NRS),
* chronic lumbosacral radicular pain lasting ≥12 weeks,
* dominant leg pain with less intense back pain,
* the previous failure of conservative management such as physiotherapy, exercise therapy, or analgesic medications.
* segmental pain of a radicular nature originating from the lumbar segments and with a shooting or lancinating quality corresponding to a dermatome suggestive of the involved nerve root.
* availability of computed tomography/magnetic resonance imaging findings of pathology concordant with the side and level of their clinical features.

Exclusion Criteria:

* patient refusal to participate in the study,
* age <18 years,
* pregnant or nursing
* pain <4-points on NRS,
* acute pain of onset lasting<12 weeks,
* progressive motor weakness in the affected leg,
* allergies to local anesthetics, contrast dyes or steroids
* significant anatomic deformity (either congenital or acquired) making it difficult to access the foramen as evidenced by computed tomography/magnetic resonance imaging
* presence of cancer accounting for back pain
* patients with platelet dysfunction, bleeding disorder or continuing anticoagulant treatment
* steroid injection within the previous 12 weeks,
* systemic infection,
* injection site infection,
* unstable medical or psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
pain scores | before the procedure and at 1, 2 and 3 months after the treatment
  Changes in pain scores, as reported by the patients via the NRS scores, will be analyzed before the procedure and at 1, 2 and 3 months after the treatment
quality of life and activities of daily living | before the procedure and at 1, 2 and 3 months after the treatment
  The potential changes in quality of life and activities of daily living will be measured by validated Roland Disability Questionnaire or Oswestry Disability Index scores

SECONDARY OUTCOMES:
adverse events | immediately and for up to 72 hours after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vadim Tashlikov, M.D., Principal Investigator — Sheba Medical Center Hospital, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howe JF, Loeser JD, Calvin WH. Mechanosensitivity of dorsal root ganglia and chronically injured axons: a physiological basis for the radicular pain of nerve root compression. Pain. 1977 Feb;3(1):25-41. doi: 10.1016/0304-3959(77)90033-1. PMID 195255
- [Background] Hildebrandt B, Wust P, Ahlers O, Dieing A, Sreenivasa G, Kerner T, Felix R, Riess H. The cellular and molecular basis of hyperthermia. Crit Rev Oncol Hematol. 2002 Jul;43(1):33-56. doi: 10.1016/s1040-8428(01)00179-2. PMID 12098606
- [Background] Koh W, Choi SS, Karm MH, Suh JH, Leem JG, Lee JD, Kim YK, Shin J. Treatment of chronic lumbosacral radicular pain using adjuvant pulsed radiofrequency: a randomized controlled study. Pain Med. 2015 Mar;16(3):432-41. doi: 10.1111/pme.12624. Epub 2014 Dec 19. PMID 25530347
- [Background] Van Boxem K, van Bilsen J, de Meij N, Herrler A, Kessels F, Van Zundert J, van Kleef M. Pulsed radiofrequency treatment adjacent to the lumbar dorsal root ganglion for the management of lumbosacral radicular syndrome: a clinical audit. Pain Med. 2011 Sep;12(9):1322-30. doi: 10.1111/j.1526-4637.2011.01202.x. Epub 2011 Aug 3. PMID 21812907
- [Background] Yonezawa M, Otsuka T, Matsui N, Tsuji H, Kato KH, Moriyama A, Kato T. Hyperthermia induces apoptosis in malignant fibrous histiocytoma cells in vitro. Int J Cancer. 1996 May 3;66(3):347-51. doi: 10.1002/(SICI)1097-0215(19960503)66:33.0.CO;2-8. PMID 8621256
- [Background] Chua NH, Vissers KC, Sluijter ME. Pulsed radiofrequency treatment in interventional pain management: mechanisms and potential indications-a review. Acta Neurochir (Wien). 2011 Apr;153(4):763-71. doi: 10.1007/s00701-010-0881-5. Epub 2010 Nov 30. PMID 21116663
- [Background] Hagiwara S, Iwasaka H, Takeshima N, Noguchi T. Mechanisms of analgesic action of pulsed radiofrequency on adjuvant-induced pain in the rat: roles of descending adrenergic and serotonergic systems. Eur J Pain. 2009 Mar;13(3):249-52. doi: 10.1016/j.ejpain.2008.04.013. Epub 2008 Jun 6. PMID 18539061
- [Background] Laboureyras E, Rivat C, Cahana A, Richebe P. Pulsed radiofrequency enhances morphine analgesia in neuropathic rats. Neuroreport. 2012 Jun 20;23(9):535-9. doi: 10.1097/WNR.0b013e3283541179. PMID 22546701
- [Background] Vallejo R, Tilley DM, Williams J, Labak S, Aliaga L, Benyamin RM. Pulsed radiofrequency modulates pain regulatory gene expression along the nociceptive pathway. Pain Physician. 2013 Sep-Oct;16(5):E601-13. PMID 24077210
- [Background] Wu B, Ni J, Zhang C, Fu P, Yue J, Yang L. Changes in spinal cord met-enkephalin levels and mechanical threshold values of pain after pulsed radio frequency in a spared nerve injury rat model. Neurol Res. 2012 May;34(4):408-14. doi: 10.1179/1743132812Y.0000000026. PMID 22643086
- [Background] 11. Sluijter ME, Cosman ER, Rittman IIWB, van Kleef M. The effects of pulsed radiofrequency field applied to the dorsal root ganglion-A preliminary report. The Pain Clinic 1998;11(2):109-17.
- [Background] Munglani R. The longer term effect of pulsed radiofrequency for neuropathic pain. Pain. 1999 Mar;80(1-2):437-9. doi: 10.1016/s0304-3959(98)00183-3. PMID 10204759
- [Background] Teixeira A, Grandinson M, Sluijter ME. Pulsed radiofrequency for radicular pain due to a herniated intervertebral disc--an initial report. Pain Pract. 2005 Jun;5(2):111-5. doi: 10.1111/j.1533-2500.2005.05207.x. PMID 17177757
- [Background] Abejon D, Garcia-del-Valle S, Fuentes ML, Gomez-Arnau JI, Reig E, van Zundert J. Pulsed radiofrequency in lumbar radicular pain: clinical effects in various etiological groups. Pain Pract. 2007 Mar;7(1):21-6. doi: 10.1111/j.1533-2500.2007.00105.x. PMID 17305674
- [Background] Simopoulos TT, Kraemer J, Nagda JV, Aner M, Bajwa ZH. Response to pulsed and continuous radiofrequency lesioning of the dorsal root ganglion and segmental nerves in patients with chronic lumbar radicular pain. Pain Physician. 2008 Mar-Apr;11(2):137-44. PMID 18354708
- [Background] Chao SC, Lee HT, Kao TH, Yang MY, Tsuei YS, Shen CC, Tsou HK. Percutaneous pulsed radiofrequency in the treatment of cervical and lumbar radicular pain. Surg Neurol. 2008 Jul;70(1):59-65; discussion 65. doi: 10.1016/j.surneu.2007.05.046. Epub 2008 Jan 22. PMID 18207554
- [Background] Shabat S, Pevsner Y, Folman Y, Gepstein R. Pulsed radiofrequency in the treatment of patients with chronic neuropathic spinal pain. Minim Invasive Neurosurg. 2006 Jun;49(3):147-9. doi: 10.1055/s-2006-944238. PMID 16921454
- [Background] Pevzner E, David R, Leitner Y, Pekarsky I, Folman Y, Gepstein R. [Pulsed radiofrequency treatment of severe radicular pain]. Harefuah. 2005 Mar;144(3):178-80, 231. Hebrew. PMID 15844456
- [Background] Leung SM, Chau WW, Law SW, Fung KY. Clinical value of transforaminal epidural steroid injection in lumbar radiculopathy. Hong Kong Med J. 2015 Oct;21(5):394-400. doi: 10.12809/hkmj144310. Epub 2015 Aug 14. PMID 26273016
- [Background] Bateman BT, Brenner GJ. An important step forward in the safe use of epidural steroid injections. Anesthesiology. 2015 May;122(5):964-6. doi: 10.1097/ALN.0000000000000615. No abstract available. PMID 25668413
- [Background] Rathmell JP, Benzon HT, Dreyfuss P, Huntoon M, Wallace M, Baker R, Riew KD, Rosenquist RW, Aprill C, Rost NS, Buvanendran A, Kreiner DS, Bogduk N, Fourney DR, Fraifeld E, Horn S, Stone J, Vorenkamp K, Lawler G, Summers J, Kloth D, O'Brien D Jr, Tutton S. Safeguards to prevent neurologic complications after epidural steroid injections: consensus opinions from a multidisciplinary working group and national organizations. Anesthesiology. 2015 May;122(5):974-84. doi: 10.1097/ALN.0000000000000614. PMID 25668411
- [Background] Racoosin JA, Seymour SM, Cascio L, Gill R. Serious Neurologic Events after Epidural Glucocorticoid Injection--The FDA's Risk Assessment. N Engl J Med. 2015 Dec 10;373(24):2299-301. doi: 10.1056/NEJMp1511754. Epub 2015 Oct 7. No abstract available. PMID 26444582
- [Background] Kennedy DJ, Levin J, Rosenquist R, Singh V, Smith C, Stojanovic MP, Vorobeychik Y. Epidural Steroid Injections are Safe and Effective: Multisociety Letter in Support of the Safety and Effectiveness of Epidural Steroid Injections. Pain Med. 2015 May;16(5):833-8. doi: 10.1111/pme.12667. Epub 2015 Jan 13. PMID 25586082
- [Background] Bhargava A, DePalma MJ, Ludwig S, Gelb D, Slipman CW. Injection therapy for lumbar radiculopathy.Curr OpinOrthop 2005;16:152-7
- [Background] Abdi S, Datta S, Trescot AM, Schultz DM, Adlaka R, Atluri SL, Smith HS, Manchikanti L. Epidural steroids in the management of chronic spinal pain: a systematic review. Pain Physician. 2007 Jan;10(1):185-212. PMID 17256030